CLINICAL TRIAL: NCT04374357
Title: Examining Prison Inmates' Attitudes and Internal Emotional States: Forgiveness, Anger, Anxiety, Depression, Hope, and Social Desirability
Brief Title: Examining Prison Inmates' Attitudes and Internal Emotional States
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Department of Corrections, State of Wisconsin (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2016-0593; A173000 (Other: University of Wisconsin, Madison); EDUC/EDUC PSYCH (Other: University of Wisconsin, Madison)
Record Dates: First submitted 2020-04-28; First posted 2020-05-05 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Forgiveness
Keywords: Forgiveness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is the first part of a two-tiered research project to propose a novel approach-forgiveness therapy-to corrections. This study is a non-intervention study and aims to demonstrate the need to introduce the concepts of forgiveness and Forgiveness Therapy within prisons. This study is focused on the extent to which men in a maximum-security prison experienced considerable injustice against them (such as in a family context as he was growing up) prior to committing serious crimes. Variables associated with this prior unjust treatment included the level of forgiveness and variables of current psychological well-being. Since this study provided the rationale and participants' matching data (eligibility) for the subsequent interventional study (Study 2, "Proposing Forgiveness Therapy in Prison") in which psychological treatments applied to the inmates, investigator refer to this study as Study 1.

DETAILED DESCRIPTION:
Current study (Study 1) consisted of 103 men in a maximum-security prison in the Midwestern United States. The research aimed to demonstrate the necessity of introducing forgiveness concepts and Forgiveness Therapy within the prison. This study collected percentage and correlational data regarding the presence of hurtful unfair treatments and psychological compromises, recognizing the style of the story-recalling (e.g. repetitive angry retelling; focus on damage; focus on fear; focus on despair, and so forth), rating of the injury types, and severity and age of occurrence. Inmates' stories were coded and analyzed by up to five researchers. The first wave of data examined a) whether participants have been treated deeply unfairly prior to their crime and imprisonment and the degree of severity; b) the degree to which the participants' show both excessive anger and unforgiveness toward those who acted unjustly as well as their expressions in crimes-direct contribution to their choice of harming the innocent; and c) the relationship among the excessive anger, forgiveness, and related emotional sufferings and psychological distresses such as anxiety and depression. Case studies were also conducted. Reliability and validation of 30-Item Enright forgiveness inventory (EFI-30) in the prison context were also tested. In general, we tested the following hypotheses:

1. Do most inmates in this maximum-security prison experience severe unfair treatment against them before their criminal perpetrations?
2. Do most inmates in this maximum-security prison have low forgiveness towards the person who deeply hurt them?
3. Do disproportional number of inmates in this maximum-security prison have clinical compromises (e.g. excessive anger, anxiety, and depression) related to their past injustice?
4. Does higher degree of anger/anxiety in inmates correlates to the less forgiving behavior towards those who hurt them in the past, prior to their crime?

Study 1 also provided participant matching data (criteria for eligible participants) for the Forgiveness Therapy experiments of subsequent interevtional study

ELIGIBILITY:
Inclusion Criteria:

* Male prison inmates, who have never participated in forgiveness therapies, were recruited voluntarily from a maximum-security prison in Wisconsin, United States.

Exclusion Criteria:

* have participated in forgiveness workshops
* are not from maximum security prison
* female; (due to the all-male prison context)
* are illiterate (cannot write their stories and finish the scales)
* have been diagnosed with cognitive disorders or cognitive function impairment
* receive one-on-one treatment with the psychologist in prison

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Prison inmates from a maximum-security prison in Wisconsin, United States.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2017-11-11 (Actual); Study Completion 2017-11-11 (Actual)

PRIMARY OUTCOMES:
Score on Patient-Reported Outcomes Measurement Information System (PROMIS) Measures of Anger | Baseline
  National Institutes of Health PROMIS Measures of Anger (five items) was used. Items are statements about the frequency of feeling angry in the past seven days. An example is "In the past 7 days, I felt like I was ready to explode." Participants need to respond to each item on a 5-point scale from "Never" to "Always." The total scores for the anger scale range from 5 to 25. The higher scores a participant rated in one scale, the angrier participant was, in contrast with those who scored lower.
Score on Patient-Reported Outcomes Measurement Information System (PROMIS) Measures of Anxiety | Baseline
  National Institutes of Health PROMIS Measures of Anxiety (seven items) was used. Items are statements about the frequency of feeling anxious in the past seven days. An example is "In the past seven days, I found it hard to focus on anything other than my anxiety." Participants need to respond to each item on a 5-point scale from "Never" to "Always." The total scores for the anxiety scale range from 5 to 35. The higher scores a participant rated in one scale, the more anxious participant was, in contrast with those who scored lower.
Score on Patient-Reported Outcomes Measurement Information System (PROMIS) Measures of Depression | Baseline
  National Institutes of Health PROMIS Measures of Depression (eight items) was used. Items are statements about the frequency of feeling depressed in the past seven days. An example is "In the past seven days, I felt like a failure." Participants need to respond to each item on a 5-point scale from "Never" to "Always." The total scores for the anxiety scale range from 5 to 40. The higher scores a participant rated in one scale, the more depressed participant was, in contrast with those who scored lower.
Score on Herth Hope Index | Baseline
  The Herth Hope Index was used as an instrument. It has 12 items and assesses optimism toward the future with questions, such as "I have a positive outlook on life"; "I believe that each day has potential". These questions assess connectedness to positive expectations for the future, inter-connectedness with other people, and inner positive expectancy. Participants responded on a 4-point scale ranging from "strongly disagree" to "strongly agree." Two items need to be reversely coded, and the total hope score ranges from 12 to 48. A higher score means more hopefulness toward the future.
Score on Enright Forgiveness Inventory | Baseline
  Enright Forgiveness Inventory Short Form (30 items) was used as a measurement of forgiveness. It includes three subscales: affect, behavior, and cognition, with 10 items in each subscale. The introductory material at the beginning asks participants to focus on the worst injustice they experienced before their first imprisonment, and to indicate the person who unfairly treated them, time to event, degree of hurt and a brief description of the experience. Then participants were asked to think about the person who hurt them and rate the 30 items on a 6-point Likert scale ranging from "strongly disagree" to "strongly agree." Half of the items are negative statements, and reverse coding is done in the data analysis. An example of the positive items is "I feel warm toward him/her," and a negative one is "Regarding this person, I disapprove of him/her." The total forgiveness scores range from 30 to 180, with each subscale scores in the range of 10 to 60. A higher score means more forgiving.
Score on Marlowe-Crowne Social Desirability Scale | Baseline
  The Marlowe-Crowne Social Desirability Scale (20-item short version) was used here to measure if a participant is "faking good" to meet the social desirability in psychological tests. It also assesses the degree to which each participant is taking this set of questionnaires seriously or not. This 20-item short version of the Marlowe-Crowne Social Desirability Scale was developed by Strahan and Gerbasi, with 20 statements using a true/false response format. An example is "I never hesitate to go out of my way to help someone in trouble." A participant gets 1 point for each "True" response and 0 point for each "False" response to 10 socially desired statements, and the reverse points to 10 not socially desired statements. Scores range from 0 to 20. A higher score represents a higher tendency of "faking good" in the test.
Score on Maltreatment and Abuse Chronology of Exposure (MACE) Scale | Baseline
  The MACE scale includes 52 items and measures retrospectively ten types of maltreatment during each year of childhood from 1 to 18 years old. The ten subscales or types of maltreatment measured include: emotional neglect, non-verbal emotional abuse, parental physical maltreatment, parental verbal abuse, peer emotional abuse, peer physical bullying, physical neglect, sexual abuse, witnessing interparental violence, and witnessing violence to siblings.
Type of Past Injustice/Unfair Treatment assessed through category 1-5 | Baseline
  After participants write their stories by the instructions and leading questions provided, these stories were coded by 3-5 independent researchers for the type of injustice: 1-physical (e.g. hitting that can damage), 2-sexual, 3-verbal (e.g. words meant to demean), 4-failure to protect or provide (emotional abuse such as constant ignoring; failure to protect the person's psychological health; physical danger to the participant such as no food or shelter or only occasional food or shelter, for example), 5-secondary (adversity towards those who are important to the person, such as the person witnessed that father beat mother). Note: Emotional abuse cuts across all of the above categories, 1-5.
Age of participant at the time of unjust treatment | Baseline
  After participants write their stories by the instructions and leading questions provided, these stories were coded by 3-5 independent researchers for the age of the injustice/unfair treatment occurred.
"Severity of Childhood Injustice" assessed on score 1-6 | Baseline
  After participants write their stories by the instructions and leading questions provided, these stories were coded by 3-5 independent researchers for the severity of childhood injustice. Childhood injustice was scored as 1-2: mild; Scored as 3-4: moderate; Scored as 5-6: severe.
"Severity of Injustice Impact on participant's future life" assessed on score 1-6 | Baseline
  After participants write their stories by the instructions and leading questions provided, these stories were coded by 3-5 independent researchers for the severity of injustice impact for their future life after the unfair treatment. Scored as 1-2: mild; Scored as 3-4: moderate; Scored as 5-6: severe.
Percentage on participants who shared the experience of injustice with anyone | Baseline
  After participants write their stories by the instructions and leading questions provided, these stories were coded by 3-5 independent researchers for whether they shared this/those experience(s) with anyone, or anyone asked before. If so, who? Investigator collected participants' answers in word and analyzed the percentage data.
Percentage on participants who seeked help after the injustice experience | Baseline
  After participants write their stories by the instructions and leading questions provided, these stories were coded by 3-5 independent researchers for whether anyone recognized/helped with healing their hurt. If so, who? Investigator collected participants' answers in word and analyzed the percentage data.

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Enright, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Columbia Correctional Institution, Portage, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Erzar T, Yu L, Enright RD, Kompan Erzar K. Childhood Victimization, Recent Injustice, Anger, and Forgiveness in a Sample of Imprisoned Male Offenders. Int J Offender Ther Comp Criminol. 2019 Jan;63(1):18-31. doi: 10.1177/0306624X18781782. Epub 2018 Jun 21. PMID 29926759
- [Background] Lee YR, Enright RD. A Forgiveness Intervention for Women With Fibromyalgia Who Were Abused in Childhood: A Pilot Study. Spiritual Clin Pract (Wash D C ). 2014 Sep;1(3):203-217. doi: 10.1037/scp0000025. Epub 2014 Aug 25. PMID 25914886
- [Background] Waltman MA, Russell DC, Coyle CT, Enright RD, Holter AC, M Swoboda C. The effects of a forgiveness intervention on patients with coronary artery disease. Psychol Health. 2009 Jan;24(1):11-27. doi: 10.1080/08870440903126371. PMID 20186637
- [Background] Hansen MJ, Enright RD, Baskin TW, Klatt J. A palliative care intervention in forgiveness therapy for elderly terminally ill cancer patients. J Palliat Care. 2009 Spring;25(1):51-60. PMID 19445342
- [Background] Reed GL, Enright RD. The effects of forgiveness therapy on depression, anxiety, and posttraumatic stress for women after spousal emotional abuse. J Consult Clin Psychol. 2006 Oct;74(5):920-9. doi: 10.1037/0022-006X.74.5.920. PMID 17032096
- [Background] Lin WF, Mack D, Enright RD, Krahn D, Baskin TW. Effects of forgiveness therapy on anger, mood, and vulnerability to substance use among inpatient substance-dependent clients. J Consult Clin Psychol. 2004 Dec;72(6):1114-21. doi: 10.1037/0022-006X.72.6.1114. PMID 15612857
- [Background] McKay KM, Hill MS, Freedman SR, Enright RD. Towards a feminist empowerment model of forgiveness psychotherapy. Psychotherapy (Chic). 2007 Mar;44(1):14-29. doi: 10.1037/0033-3204.44.1.14. PMID 22122165
- [Background] Yu, L., Gambaro, M., Komoski, M. C., Song, M. J., Song, M., Teslik, M., Wollner, B., & Enright, R. D. (2018). The Silent Injustices against Men in Maximum Security Prison and the Need for Forgiveness Therapy: Two Case Studies. Journal of Forensic Psychology, 3, 137. DOI: 10.4172/2475-319X.1000137.
- [Background] Enright, R. D., Erzar, T., Gambaro, M., Komoski, M. C., O'Boyle, J., Reed, G., & ... Yu, L. (2016). Proposing Forgiveness Therapy for those in Prison: An Intervention Strategy for Reducing Anger and Promoting Psychological Health. Journal of Forensic Psychology, 1, 116. DOI: 10.4172/2475-319X.1000116.
- See also: Project descriptions on this study — https://www.researchgate.net/project/Proposing-Forgiveness-Therapy-for-Those-in-Prison-An-Intervention-for-Reducing-Anger-and-Promoting-Psychological-Health